CLINICAL TRIAL: NCT04340011
Title: Colposcopy Education Using Operant Learning
Acronym: Colpo
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Sponsor
Other Study IDs: 22034
Record Dates: First submitted 2020-01-13; First posted 2020-04-09 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Educational Problems; Cervix, Dysplasia
Keywords: colposcopy; resident education
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Colposcopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Colposcopy — prospective resident education for colposcopy
  Other Names: prospective resident education

SUMMARY:
Images will be collected during routine colposcopy and paired with their pathology results to be used for resident education

DETAILED DESCRIPTION:
Identifying information will be removed and operant learning techniques will be applied to better educate residents on colposcopy.

ELIGIBILITY:
Inclusion Criteria:

* ability to give informed consent
* age 21or older
* undergoing clinically indicated colposcopy

Exclusion Criteria:

* under 21 years of age

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — colposcopy only performed in female population
Study Population: Females over the age of 21 undergoing clinically indicated coposcopy that are able to give informed consent
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Resident accuracy in identifying sites for biopsy during Colposcopy | 1 year
  using colposcopic images obtained during routine patient care residents will complete quiz from images with immediate results of the test to assess the accuracy of visual cues to biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Cantrell, MD, Principal Investigator — University of Virginia
Locations (1):
- Univeristy of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Once pathology is confirmed 3-4 weeks post colposcopy all PHI will be removed from the participant